CLINICAL TRIAL: NCT06674928
Title: Developmental Trajectory of Gene and Life Participation in Children With Developmental Delay
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301017A3
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-10

CONDITIONS: Genetics; Life Participation
Keywords: Developmental delay; Life participation; Quality of life; Whole-exome sequencing; Gene; Children Development
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Developing Children: Children that were satisfied with the criteria as average or "on-time" growth based on the attainment of specific physical, cognitive, linguistic, social-emotional, and behavioral milestones across specific stages.
- Developmental Delay Children: Children who has not gained the developmental skills expected of him or her, compared to others of the same age.

SUMMARY:
The goal of this observational study is to learn the factors affecting the quality of life in children's development.

The main hypothesis for this study is:

If the level of well-being increases in age, could the quality of life be enhanced in terms of function and participation?

Participant will be given assessment every year for five years in total. No intervention will be given during the whole study period.

ELIGIBILITY:
Normal developing children

Inclusion Criteria:

* Agreeing in consent
* In the age range of 6-15 years old

Exclusion Criteria:

* Diseases of Central Nervous System
* Diseases of Neuromuscular
* Nature deficit disorder
* Genetic Disorder
* Sensory Integration disorder
* Auditory disorder

Development delay children

Inclusion Criteria:

* Agreeing in consent
* In the age range of 6-15 years old
* Diagnosed of Developmental Delay

Exclusion Criteria:

* Diseases of Central Nervous System
* Diseases of Neuromuscular
* Nature deficit disorder
* Genetic Disorder
* Sensory Integration disorder
* Auditory disorder

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Control and experimental group
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Score of participation (< 3y) | baseline
  Children Assessment of Participation and Enjoyment and Preferences for Activity of Children (Higher scores means a better outcome.)
Score of participation (3y > 15y) | Baseline
  Pediatric Quality of Life Inventory TM (Scores from 0 to 102, higher scores mean a better outcome.)

SECONDARY OUTCOMES:
Gene Test | Baseline
  Whole-Exome Sequencing (Use Burrows-Wheeler Aligner (BWA) 85, Samtools86, Picard, Genome Analysis Toolkit (GATK) to screen out the variant discovery and genotyping.)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD,PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan